CLINICAL TRIAL: NCT02267811
Title: The Effect of OrthoPulse™ on the Rate of Orthodontic Tooth Movement During Alignment With Fixed Appliances
Brief Title: The Effect of OrthoPulse™ on the Rate of Orthodontic Tooth Movement
Acronym: BX8RN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX8RN
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Malocclusion
Keywords: Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™
MeSH Terms: conditions — Malocclusion | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fixed Orthodontic Treatment with OrthoPulse™ (Experimental): Subjects assigned to this group receive orthodontic treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Interventions: Other: Orthodontic Treatment; Device: OrthoPulse™
- Fixed Orthodontic Treatment (Experimental): Subjects assigned to this group receive orthodontic treatment with no OrthoPulse™ treatment.
  Interventions: Other: Orthodontic Treatment

INTERVENTIONS:
Other: Orthodontic Treatment — Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Device: OrthoPulse™ — Participants carry out daily OrthoPulse™ treatments at home.
  Arms: Fixed Orthodontic Treatment with OrthoPulse™

SUMMARY:
This open label study is designed to evaluate the ability of OrthoPulse™ to safely and effectively increase the rate of orthodontic tooth movement with fixed appliances.

DETAILED DESCRIPTION:
The primary aim of this study is to determine if daily OrthoPulse™ use affects the rate of orthodontic tooth movement during alignment with fixed appliances in the mandibular arch.

The secondary aim of this study is to determine whether patients treated with OrthoPulse demonstrate root resorption beyond what is commonly expected during orthodontic treatment.

The study also aims to collect confirmatory evidence on the safety of the device.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and scheduled for full mouth fixed orthodontic treatment
* Moderate to severe crowding (LII ≥ 3 mm), with no labio-lingually displaced teeth
* Class I or Class II by 1/2 cusp or less
* Non-extraction in both arches
* Age 11- 60
* Good oral hygiene
* Non-smokerInclud

Exclusion Criteria:

* Pregnant females
* Patient is currently enrolled in another clinical study
* Patient decided on Invisalign® rather than braces
* Periodontally involved teeth
* Use of bisphosphonates (osteoporosis drugs) during the study
* Patient plans to move over the treatment period
* Spaces between anterior teeth

Ages: 11 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brawn, DDS, Study Director — Biolux Research
Locations (1):
- Stone Oak Orthodontics, San Antonio, Texas, United States

REFERENCES:
- [Background] Skidmore KJ, Brook KJ, Thomson WM, Harding WJ. Factors influencing treatment time in orthodontic patients. Am J Orthod Dentofacial Orthop. 2006 Feb;129(2):230-8. doi: 10.1016/j.ajodo.2005.10.003. PMID 16473715
- [Background] Kawakami M, Takano-Yamamoto T. Local injection of 1,25-dihydroxyvitamin D3 enhanced bone formation for tooth stabilization after experimental tooth movement in rats. J Bone Miner Metab. 2004;22(6):541-6. doi: 10.1007/s00774-004-0521-3. PMID 15490263
- [Background] Yamasaki K, Shibata Y, Imai S, Tani Y, Shibasaki Y, Fukuhara T. Clinical application of prostaglandin E1 (PGE1) upon orthodontic tooth movement. Am J Orthod. 1984 Jun;85(6):508-18. doi: 10.1016/0002-9416(84)90091-5. PMID 6587784
- [Background] Seifi M, Eslami B, Saffar AS. The effect of prostaglandin E2 and calcium gluconate on orthodontic tooth movement and root resorption in rats. Eur J Orthod. 2003 Apr;25(2):199-204. doi: 10.1093/ejo/25.2.199. PMID 12737218
- [Background] Hashimoto F, Kobayashi Y, Mataki S, Kobayashi K, Kato Y, Sakai H. Administration of osteocalcin accelerates orthodontic tooth movement induced by a closed coil spring in rats. Eur J Orthod. 2001 Oct;23(5):535-45. doi: 10.1093/ejo/23.5.535. PMID 11668873
- [Background] Madan MS, Liu ZJ, Gu GM, King GJ. Effects of human relaxin on orthodontic tooth movement and periodontal ligaments in rats. Am J Orthod Dentofacial Orthop. 2007 Jan;131(1):8.e1-10. doi: 10.1016/j.ajodo.2006.06.014. PMID 17208099
- [Background] Frost HM. Wolff's Law and bone's structural adaptations to mechanical usage: an overview for clinicians. Angle Orthod. 1994;64(3):175-88. doi: 10.1043/0003-3219(1994)0642.0.CO;2. PMID 8060014
- [Background] Davidovitch Z, Finkelson MD, Steigman S, Shanfeld JL, Montgomery PC, Korostoff E. Electric currents, bone remodeling, and orthodontic tooth movement. I. The effect of electric currents on periodontal cyclic nucleotides. Am J Orthod. 1980 Jan;77(1):14-32. doi: 10.1016/0002-9416(80)90221-3. PMID 6243447
- [Background] Nishimura M, Chiba M, Ohashi T, Sato M, Shimizu Y, Igarashi K, Mitani H. Periodontal tissue activation by vibration: intermittent stimulation by resonance vibration accelerates experimental tooth movement in rats. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4):572-83. doi: 10.1016/j.ajodo.2006.01.046. PMID 18405822
- [Background] Bernabe E, Flores-Mir C. Estimating arch length discrepancy through Little's Irregularity Index for epidemiological use. Eur J Orthod. 2006 Jun;28(3):269-73. doi: 10.1093/ejo/cji112. Epub 2006 Apr 28. PMID 16648212
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Limpanichkul W, Godfrey K, Srisuk N, Rattanayatikul C. Effects of low-level laser therapy on the rate of orthodontic tooth movement. Orthod Craniofac Res. 2006 Feb;9(1):38-43. doi: 10.1111/j.1601-6343.2006.00338.x. PMID 16420273
- [Background] Almasoud N, Bearn D. Little's irregularity index: photographic assessment vs study model assessment. Am J Orthod Dentofacial Orthop. 2010 Dec;138(6):787-94. doi: 10.1016/j.ajodo.2009.01.031. PMID 21130338
- [Background] Tran AM, Rugh JD, Chacon JA, Hatch JP. Reliability and validity of a computer-based Little irregularity index. Am J Orthod Dentofacial Orthop. 2003 Mar;123(3):349-51. doi: 10.1067/mod.2003.76. No abstract available. PMID 12637908
- [Background] Canuto LF, de Freitas MR, de Freitas KM, Cancado RH, Neves LS. Long-term stability of maxillary anterior alignment in non-extraction cases. Dental Press J Orthod. 2013 May-Jun;18(3):46-53. doi: 10.1590/s2176-94512013000300009. PMID 24094011
- [Background] Krieger E, Drechsler T, Schmidtmann I, Jacobs C, Haag S, Wehrbein H. Apical root resorption during orthodontic treatment with aligners? A retrospective radiometric study. Head Face Med. 2013 Aug 14;9:21. doi: 10.1186/1746-160X-9-21. PMID 23941626
- [Background] Fritz U, Diedrich P, Wiechmann D. Apical root resorption after lingual orthodontic therapy. J Orofac Orthop. 2003 Nov;64(6):434-42. doi: 10.1007/s00056-003-0243-5. English, German. PMID 14628135
- [Background] Bergius M, Berggren U, Kiliaridis S. Experience of pain during an orthodontic procedure. Eur J Oral Sci. 2002 Apr;110(2):92-8. doi: 10.1034/j.1600-0722.2002.11193.x. PMID 12013568
- [Background] Erdinc AM, Dincer B. Perception of pain during orthodontic treatment with fixed appliances. Eur J Orthod. 2004 Feb;26(1):79-85. doi: 10.1093/ejo/26.1.79. PMID 14994886
- [Background] Jones M, Chan C. The pain and discomfort experienced during orthodontic treatment: a randomized controlled clinical trial of two initial aligning arch wires. Am J Orthod Dentofacial Orthop. 1992 Oct;102(4):373-81. doi: 10.1016/0889-5406(92)70054-e. PMID 1456222
- [Background] Liu Z, McGrath C, Hagg U. Changes in oral health-related quality of life during fixed orthodontic appliance therapy: an 18-month prospective longitudinal study. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):214-9. doi: 10.1016/j.ajodo.2009.08.029. PMID 21300250
- [Background] Zhang M, McGrath C, Hagg U. Changes in oral health-related quality of life during fixed orthodontic appliance therapy. Am J Orthod Dentofacial Orthop. 2008 Jan;133(1):25-9. doi: 10.1016/j.ajodo.2007.01.024. PMID 18174067
- [Background] Bernabe E, Sheiham A, Tsakos G, Messias de Oliveira C. The impact of orthodontic treatment on the quality of life in adolescents: a case-control study. Eur J Orthod. 2008 Oct;30(5):515-20. doi: 10.1093/ejo/cjn026. Epub 2008 Aug 27. PMID 18753305
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Linge BO, Linge L. Apical root resorption in upper anterior teeth. Eur J Orthod. 1983 Aug;5(3):173-83. doi: 10.1093/ejo/5.3.173. No abstract available. PMID 6578039
- [Background] Lund H, Grondahl K, Hansen K, Grondahl HG. Apical root resorption during orthodontic treatment. A prospective study using cone beam CT. Angle Orthod. 2012 May;82(3):480-7. doi: 10.2319/061311-390.1. Epub 2011 Sep 16. PMID 21919826
- [Background] Makedonas D, Lund H, Hansen K. Root resorption diagnosed with cone beam computed tomography after 6 months and at the end of orthodontic treatment with fixed appliances. Angle Orthod. 2013 May;83(3):389-93. doi: 10.2319/042012-332.1. Epub 2012 Oct 23. PMID 23092202
- [Background] Heritier SR, Gebski VJ, Keech AC. Inclusion of patients in clinical trial analysis: the intention-to-treat principle. Med J Aust. 2003 Oct 20;179(8):438-40. doi: 10.5694/j.1326-5377.2003.tb05627.x. No abstract available. PMID 14558871
- [Background] Wright N, Modarai F, Cobourne MT, Dibiase AT. Do you do Damon(R)? What is the current evidence base underlying the philosophy of this appliance system? J Orthod. 2011 Sep;38(3):222-30. doi: 10.1179/14653121141479. PMID 21875995
- [Background] Celar A, Schedlberger M, Dorfler P, Bertl M. Systematic review on self-ligating vs. conventional brackets: initial pain, number of visits, treatment time. J Orofac Orthop. 2013 Jan;74(1):40-51. doi: 10.1007/s00056-012-0116-x. Epub 2013 Jan 10. PMID 23299650

RESULTS

PARTICIPANT FLOW:
Groups:
- BX8RN: Orthodontic Treatment With OrthoPulse™ (Treatment): Subjects assigned to this group receive orthodontic treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- BX8RN: Orthodontic Treatment (Control): Subjects assigned to this group receive orthodontic treatment without OrthoPulse™ treatment.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Period: Overall Study
Arm/Group | BX8RN: Orthodontic Treatment With OrthoPulse™ (Treatment) | BX8RN: Orthodontic Treatment (Control)
Started | 16 | 17
Completed | 15 | 15
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- BX8RN: OrthoPulse™ (Treatment): Subjects assigned to this group receive orthodontic treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- BX8RN: Orthodontic Treatment With no OrthoPulse™ (Control): Subjects assigned to this group receive orthodontic treatment with no daily OrthoPulse™ treatments.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
- Total: Total of all reporting groups
Arm/Group | BX8RN: OrthoPulse™ (Treatment) | BX8RN: Orthodontic Treatment With no OrthoPulse™ (Control) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 4 | 11 | 15
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Whether OrthoPulse Use Affects the Rate of Orthodontic Tooth Movement During Full Mouth Fixed Orthodontic Treatment
Description: Rate of participants orthodontic tooth movement using Little's Index of Irregularity (LII) measured in millimeters per week during alignment.
Time Frame: Participants will be followed for the duration of their orthodontic treatment, an expected average of 1-2 years, depending on the severity of the case.
Measure: Mean (Standard Deviation); unit: millimeters per week
Arm/Group | BX8RN: Orthodontic Treatment With OrthoPulse™ (Treatment) | BX8RN: Orthodontic Treatment (Control)
Number analyzed (Participants) | 15 | 15
millimeters per week | 1.09 (.68) | .39 (.14)

2. Secondary Outcome: Safety Evidence of OrthoPulse™ Use
Description: The number of significant adverse events reported from time of participant enrolment to study completion for all study participants
Time Frame: as for outcome 1
Measure: Number; unit: Adverse Events
Groups:
- Fixed Orthodontic Treatment With OrthoPulse™ (Treatment): Subjects assigned to this group receive orthodontic treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- Fixed Orthodontic Treatment (Control): Subjects assigned to this group receive orthodontic treatment with no OrthoPulse™ treatment.
  Orthodontic Treatment: Patients are treated for orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Arm/Group | Fixed Orthodontic Treatment With OrthoPulse™ (Treatment) | Fixed Orthodontic Treatment (Control)
Number analyzed (Participants) | 15 | 15
Adverse Events | 0 | 0

3. Secondary Outcome: Degree of External Apical Root Resorption (EARR)
Description: The amount of EARR experienced as assessed at six (6) months or later after starting treatment. External Apical Root Resorption can result from orthodontic tooth movement. External apical root resorption is the shortening of the root and affects root surface(s), which can result in loss of tooth structure. External apical root resorption is being determined in this study by comparing root lengths from initial to six (6) months or later after starting treatment. The measurements are taken from the crown to the root apex in millimeters.
  A positive number under the measure of dispersion signifies root resorption.
Time Frame: Assessed at six (6) months or later after starting treatment, up to two (2) years.
Population: The overall number of participants is not consistent with the number of participants analyzed in this arm because the panoramic radiographs required to analyze the EARR were not available for the remaining 11 participants.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Fixed Orthodontic Treatment With OrthoPulse™ (Treatment) | Fixed Orthodontic Treatment (Control)
Number analyzed (Participants) | 10 | 9
millimeters | 0.02 (.86) | -0.11 (.87)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at all visits from the time of participant enrolment through the study final visit, two (2) years or less.
Description: The definitions for adverse event and/or serious adverse event used in this study do not differ from ClinicalTrials.gov.
Arm/Group | Fixed Orthodontic Treatment With OrthoPulse™ (Treatment) | Fixed Orthodontic Treatment (Control)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No